CLINICAL TRIAL: NCT06403436
Title: A Phase 1, First-in-Human, Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of TT125-802 in Subjects With Advanced Solid Tumors
Brief Title: A Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of TT125-802 in Subjects With Advanced Solid Tumors
Acronym: TT-CSP-001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TOLREMO therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT-CSP-001
Record Dates: First submitted 2024-04-12; First posted 2024-05-07 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; Adult Solid Tumor; Adult Disease; Cancer; NSCLC; EGFR; KRAS G12C; Squamous Cell Lung Cancer
Keywords: TOLREMO; Drug resistance; TT125-802; Small molecule; Bromodomain inhibitor; NSCLC
MeSH Terms: conditions — Disease; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TT125-802 single agent (Experimental)
  Interventions: Drug: TT125-802

INTERVENTIONS:
Drug: TT125-802 — TT125-802 administered orally

SUMMARY:
The purpose of this study is to test the safety and therapeutic effect of TT125-802 (single agent) in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
The purpose of this Phase 1, First-in-Human, Open-label Study is to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of TT125-802 as single agent in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Males and nonpregnant and non-breastfeeding females, aged ≥ 18 years of age at the time of signing the informed consent.
* Subjects with advanced solid tumors resistant or refractory to standard treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Measurable disease per RECIST 1.1 criteria.
* Adequate hematological function defined by absolute neutrophil count, ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L, and hemoglobin ≥ 9 g/dL, and without growth factor treatment or blood transfusion within 2 weeks before the study intervention start.
* Adequate hepatic function defined by total bilirubin level ≤ 1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) level ≤ 3 × ULN, and an alanine aminotransferase (ALT) level ≤ 3 × ULN.
* Adequate renal function defined by creatinine clearance > 60 mL/min according to the Cockcroft-Gault equation or creatinine levels <1.5 mg/dl.
* Adequate coagulation laboratory assessments, as follows: Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x upper limit of normal (ULN), or international normalized ratio (INR) < 1.5 or within target range if on prophylactic anticoagulation therapy.
* Life expectancy of > 3 months, in the opinion of the Investigator.
* Willing to adhere to contraception, egg and sperm donation, the fasting requirement, and other criteria as described in lifestyle restrictions
* Capable of giving signed informed consent.

Exclusion Criteria:

* Clinically significant (i.e., active) uncontrolled intercurrent illness.
* Presence of brain metastases unless clinically stable.
* History or presence of malignancies unless curatively treated with no evidence of disease ≥ 2 years.
* Subjects with known human immunodeficiency virus and/or active viral hepatitis (B and/or C), and subjects on viral hepatitis B therapy are excluded. However, subjects with hepatitis C treated with curative therapy are not considered actively infected.
* Subject received a live vaccine within 30 days prior to the first dose of the study treatment administration.
* Serious gastrointestinal bleeding within 3 months, refractory nausea and vomiting, uncontrolled diarrhea, known malabsorption, significant small bowel resection or gastric bypass surgery, use of feeding tubes, other chronic gastrointestinal disease, and/or other situation that may preclude adequate absorption of oral medications.
* Subjects that have received a strong CYP3A4 inhibitor within 7 days prior to the first dose of TT125-802 or a strong CYP3A4 inducer within 14 days prior to the first dose of TT125-802.
* Hypersensitivity to the active substance or to any of the excipients of TT125-802.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (AEs) and serious adverse events (SAEs) | Day 1 to approximately 16 weeks
Frequency of dose interruptions and dose reductions | Day 1 to approximately 16 weeks
Incidence of dose-limiting toxicities (DLTs) | Day 1 to Day 21
Recommended Dose(s) for Expansion | Day 1 to Day 21

SECONDARY OUTCOMES:
Plasma concentration of TT125-802 in blood | Day 1 to approximately 16 weeks
Objective response rate (ORR) assessed by RECIST v1.1 | Day 1 to approximately 16 weeks
Duration of response (DOR) according to RECIST v1.1 | Day 1 to approximately 16 weeks
Progression-free survival (PFS) according to RECIST v1.1 | Day 1 to approximately 16 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (2):
  - Sarah Cannon Research Institute Oncology Partners, Nashville, Tennessee
  - NEXT Oncology Virginia, Fairfax, Virginia
- Spain (3):
  - NEXT Oncology Barcelona, Barcelona
  - Vall d'Hebron Institute of Oncology, Barcelona
  - NEXT Oncology Madrid, Madrid
- Switzerland (2):
  - Ente Ospedaliero Cantonale, Bellinzona
  - Centre Hospitalier Universitaire Vaudois, Lausanne

IPD SHARING:
Plan to Share IPD: No